CLINICAL TRIAL: NCT05732337
Title: Prospective, Open Clinical Investigation to Evaluate the Effectiveness and Safety of a Topical Medical Device for the Treatment of Chickenpox Symptoms
Brief Title: Open Clinical Investigation to Evaluate the Effectiveness and Safety of a Topical Medical Device.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karo Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22E3464/ PXC_001
Record Dates: First submitted 2023-01-27; First posted 2023-02-17 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-01

CONDITIONS: Chickenpox
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Intervention Model Description: To determine the efficacy of PoxClin® CoolMousse in relieving itching associated with chickenpox after 3 days of use (using 5-point scale)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Poxclin Coolmousse (Other): A cooling mousse for application to the skin supplied in a 100 mL plastic bottle with a pump (a foamer)
  Interventions: Device: Poxclin Coolmousse

INTERVENTIONS:
Device: Poxclin Coolmousse — cooling mousse for application in the skin

SUMMARY:
The primary endpoint is the change of the itching score after 3 days of the product use in comparison to the basal value.

ELIGIBILITY:
Inclusion Criteria:

1. Female and/or male
2. Aged between 12 months to 11 years
3. phototype: I to IV
4. Subject or parent(s)/legal representative(s) must be registered with health social security or health social insurance.
5. Parent(s)/legal representative(s) having signed their written Informed Consent form (ICF) for their children's participation in the study
6. Subject and / or parent(s)/legal representative(s) able to understand the language used in the investigation centre and the information given
7. Subject or parent(s)/legal representative(s) able to comply with the protocol, follow protocol's constraints and specific requirements and able to follow the medical recommendation regarding the pathology and its requirements (treatment, social eviction etc)
8. Subjects presenting non severe and non complicated chicken pox

Exclusion Criteria:

1. Subject or parent(s)/legal representative(s) who is (are) unable to understand the information (for linguistic or psychiatric reasons) and to give his/her (their) consent to his/ her (their child) participation
2. Subject taking part or planning to participate in another clinical trial during the study in the same or another investigation centre
3. Subject or parent(s)/legal representative(s) deprived of freedom by administrative or legal decision or under guardianship
4. Subject or parent(s)/legal representative(s) admitted in a sanitary or social facility
5. Subjects planning a hospitalization during the study
6. Severe or complicated chicken pox (surinfection, profuse eruption, pneumonia, etc)
7. Having an acute, chronic, or progressive disease or dermatological condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
8. Having personal medical history liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
9. Being under any treatment for a severe or complicated chicken pox considered by the Investigator liable to interfere with the study data or incompatible with the study requirements (antiviral (Herviran) or antibiotics...)
10. Having taken any previous treatment considered by the Investigator liable to interfere with the study data or incompatible with the study requirements
11. Systemic antibiotics within 1 week before the inclusion or required during the study
12. Systemic immunosuppressive treatment within 6 months before the inclusion or required during the study

Ages: 12 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
The efficacy of PoxClin® CoolMousse in relieving itching associated with chickenpox (using 5-point scale,"none (0)" to "severe (4)" ) will be evaluated after 3 days. | 3 days
  Children should be diagnosed with chickenpox.

SECONDARY OUTCOMES:
The efficacy of the PoxClin® CoolMousse in relieving itch during chickenpox (using 5 point scale, "none (0)" to "severe (4)"): itching) will be evaluated after 7 days. | 7 days
  Children should be diagnosed with chickenpox.

CONTACTS AND LOCATIONS:
Locations (1):
- Ewa Karamon, private practice, Malbork, Poland

IPD SHARING:
Plan to Share IPD: No